CLINICAL TRIAL: NCT04989244
Title: Weight Loss Program in Infertile PCOS Women With Obesity
Brief Title: Infertile Polycystic Ovary Syndrome (PCOS) Women With Obesity and Lifestyle Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Slovenian Research Agency (Other)
Responsible Party: Principal Investigator, Tanja Burnik Papler, Assist. Prof., University Medical Centre Ljubljana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TBP1
Record Dates: First submitted 2021-07-01; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Weight Reduction Programs

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Weight loss program — Women with obesity were included to the weight loss program which included physical exercise and dietary guidelines

SUMMARY:
Infertile PCOS women with obesity were included into lifestyle change weight loss program prior to inclusion to IVF procedures. They attended group as well as individual workouts and they were advised on healthy eating.

DETAILED DESCRIPTION:
The weight loss program will consist of dietary change and exercise program which will be performed 3 times weekly.

ELIGIBILITY:
Inclusion Criteria:

* BMI over 30 kg/m2
* PCOS
* Primary or secondary infertility
* normal partner's semen

Exclusion Criteria:

* Other identifiable causes of infertility

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Body weight (kg) | 8 weeks
  Body weight before and after the weight loss program will be measured.
BMI (kg/m2) | 8 weeks
  BMI before and after the weight loss program will be calculated).
Waist circumference (cm) | 8 weeks
  Waist circumference before and after the weight loss program will be measured.
Abdominal circumference (cm) | 8 weeks
  Abdominal circumference

SECONDARY OUTCOMES:
Spontaneous conception rate | 3 months
  Spontaneous pregnancy rate after weight loss program will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of gynecology, Department of human reproduction, Ljubljana, Slovenia

REFERENCES:
- [Derived] Abdulkhalikova D, Sustarsic A, Vrtacnik Bokal E, Jancar N, Jensterle M, Burnik Papler T. The Lifestyle Modifications and Endometrial Proteome Changes of Women With Polycystic Ovary Syndrome and Obesity. Front Endocrinol (Lausanne). 2022 Jun 22;13:888460. doi: 10.3389/fendo.2022.888460. eCollection 2022. PMID 35813634